CLINICAL TRIAL: NCT00192803
Title: ACE/ACE2 Ratio in Diabetic Patients Treated With Antihypertensive Drugs
Brief Title: Non-Insulin Dependent Diabetes Mellitus (NIDDM) and Angiotensin Converting Enzyme 2 (ACE2): Diabetic Patients Treated With Antihypertensive Drugs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: ACE2.CTIL
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2006-02-23 (Estimated); Status verified 2005-09

CONDITIONS: NIDDM
Keywords: niddm; ace2; NIDDM patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — candesartan

INTERVENTIONS:
Drug: candesartan

SUMMARY:
This feasibility study is designed to examine modulation of the relative activities of ACE and ACE2 in diabetic patients following treatment with the angiotensin type 1 receptor (AT1R) antagonist, Candesartan.

This study will provide a closer insight to the possible involvement of the renin-angiotensin system (RAS)-related enzymatic components in development or attenuation of vascular pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Non-smokers
* Type II DM diagnosed patients
* Blood pressure < 135/90
* Serum HbA1C > 7%
* Serum creatinine < 1mg%
* Urine microalbumin < 300 mg/day
* Body mass index (BMI) < 35 kg/m2

Exclusion Criteria:

* Insulin-dependent diabetic patients
* Patient with persistent microalbuminuria
* Patient with history of severe hypertension
* Congestive heart failure
* Patient receiving renin-angiotensin-aldosterone system (RAAS)-related anti-hypertensive medications.
* Patient with major hepatic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20

PRIMARY OUTCOMES:
ACE and ACE2 activities in monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Keidar, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Internal Ward "A", Rambam Medical Center, Haifa, Israel